CLINICAL TRIAL: NCT00109785
Title: Positron Emitter I-124-Iododeoxyuridine to Follow DNA Metabolism on Scans and in Tumor Samples in Advanced Breast Cancer: Comparison to 18-F-2-Fluoro-2-Deoxy-(D)-Glucose, as a Tracer for Glycolysis
Brief Title: PET Scans in Patients With Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSKCC-97046; CDR0000065706 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1308
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

ARMS (1):
- PET Scans (Experimental): The first group of positron emission tomography (PET) scans is performed within 2 weeks before the first dose of chemotherapy. The second group of PET scans occur no more than 7 weeks after chemotherapy and prior to local therapy, either surgery or radiation therapy. The PET scan before initiation of chemotherapy consists of 4 imaging sessions. There is one iodine I-124 iododeoxyuridine (IUdR) PET scan (3 imaging sessions) at 1, 4-8, and 24 hours after IUdR infusion, followed by one fludeoxyglucose (FDG) PET scan (1 imaging session) 45 minutes after FDG infusion.
  Interventions: Procedure: positron emission tomography; Radiation: fludeoxyglucose F 18; Radiation: iodine I 124 iododeoxyuridine

INTERVENTIONS:
Procedure: positron emission tomography
Radiation: fludeoxyglucose F 18
Radiation: iodine I 124 iododeoxyuridine

SUMMARY:
RATIONALE: Imaging procedures such as PET scans may improve the ability to monitor the effectiveness of chemotherapy for locally advanced breast cancer.

PURPOSE: This clinical trial is studying how well PET scans work in patients with locally advanced breast cancer who will undergo chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the biologic activity of locally advanced breast cancer as measured by retention of iodine I 124 iododeoxyuridine (IUdR) on positron emission tomography (PET) scans pre- and postchemotherapy is different between patients whose tumor shrinks after treatment in comparison to patients whose tumor is stable or continues to grow.
* Demonstrate that incorporation of IUdR into tumor is in the tumor DNA at 24-36 hours post injection, as documented by tissue analysis and immunohistochemistry and that this correlates with the subsequent change in tumor dimension and proliferative activity of the tumor.
* Compare the pre and post treatment results of fludeoxyglucose (FDG) PET scanning and IUdR PET scanning in the same breast lesions as a basis for assessment of the relative metabolic change during chemotherapy.
* Further assess the biologic activity of metastatic tumor sites and their changes in size following chemotherapy to standard parameters that are used to evaluate change in tumor size, obtained under clinical standard of care for breast cancer, which will include CT scans as well as bone scans.
* Assess the accuracy of noninvasive measurement of PET measurement of the left ventricular cardiac chamber clearance of radioactivity as a substitute for arterial plasma sampling for determining metabolic rates of FDG and IUdR uptake into tumors.
* Evaluate metabolic changes in tumors as they are affected by specific chemotherapy in comparison to changes in tumor dimensions.

OUTLINE: For this study, the chemotherapy administered for an individual patient is at the discretion of the patient's primary attending physician. After chemotherapy, the patient is evaluated for surgical resection of the tumor. If the tumor is unresectable, the patient may be offered radiation therapy.

The first group of positron emission tomography (PET) scans is performed within 2 weeks before the first dose of chemotherapy. The second group of PET scans occur no more than 7 weeks after chemotherapy and prior to local therapy, either surgery or radiation therapy.

The PET scan before initiation of chemotherapy consists of 4 imaging sessions. There is one iodine I-124 iododeoxyuridine (IUdR) PET scan (3 imaging sessions) at 1, 4-8, and 24 hours after IUdR infusion, followed by one fludeoxyglucose (FDG) PET scan (1 imaging session) 45 minutes after FDG infusion.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced breast carcinoma

  * Stage T3 T4, N2 or N3 disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No history of psychiatric illness that would preclude giving informed consent
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1997-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Ann Gilewski, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States